CLINICAL TRIAL: NCT02512549
Title: 'Effects of Structured Outpatient Pulmonary Rehabilitation Intervention on Exercise Capacity and Quality of Life in Patients With Severe Chronic Obstructive Pulmonary Disease: A Randomized Controlled Study'
Brief Title: A Trial to Study the Effects of Pulmonary Rehabilitation Program on Exercise Capacity and Quality of Life in Patients With Severe Form of Chronic Obstructive Pulmonary Disease (COPD)
Acronym: RehabCOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Raju Prasad Pangeni, DM Senior Resident, Department of Pulmonary Medicine and Sleep Disorders, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AIIMS-DM Thesis
Record Dates: First submitted 2015-07-28; First posted 2015-07-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Rehabilitation
Keywords: Chronic Obstructive Pulmonary Disease; rehabiltation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehabilitation (Active Comparator): Patients with diagnosed Chronic Obstructive Pulmonary Disease with severe airflow obstruction (spirometric forced expiratory volume in one second (FEV1) below 50% of the normal) and modified medical research council (mMRC) dyspnea grading 1 to 3 will undergo pulmonary rehabilitation program thrice a week for 2 months.
  Interventions: Other: Pulmonary Rehabilitation
- Usual Care (No Intervention): Patients with COPD as described in rehabilitation arm, will be provided usual care from the hospital outpatient clinic.

INTERVENTIONS:
Other: Pulmonary Rehabilitation
  Arms: Rehabilitation

SUMMARY:
This study is a randomized parallel group controlled trial which aims to study the effects of pulmonary rehabilitation intervention on exercise capacity and quality of life in patients with severe COPD as compared to standard medical care. The expected duration is one and a half years with effect from 1st July, 2015 and will include 80 patients, 40 in each arm.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease ranks among the top five causes of unnatural deaths in India and its prevalence continues to increase. Widespread habit of smoking and the use of biomass fuels have led to such a high prevalence of COPD. The loss of physical capacity and the adverse psychosocial effects of the disorder contribute greatly to morbidity and mortality. Medicines have a limited role in improving the lung functions and physical capacity in patients with COPD. Pulmonary rehabilitation (PR) aims to return the patient with chronic obstructive pulmonary disease (COPD) to the highest level of independent functioning. This is achieved by providing individually tailored exercise training schedules, education and psychosocial support.

Pulmonary Rehabilitation has been defined by the American and the European Thoracic Societies as "a comprehensive intervention based on a thorough patient assessment followed by patient tailored therapies that include, but are not limited to, exercise training, education, and behavior change, designed to improve the physical and psychological condition of people with chronic respiratory disease and to promote the long-term adherence to health-enhancing behaviors." COPD is now considered a multi-systemic disease with frequent co-morbidities and hence the optimal management of this complex group of patients requires integrated care principles, pulmonary rehabilitation being the core component.

Patients with chronic obstructive pulmonary disease (COPD) often decrease their physical activity because exercise can worsen dyspnea. The progressive deconditioning associated with inactivity initiates a vicious cycle, with dyspnea becoming problematic at ever lower physical demands. Pulmonary rehabilitation aims to break the cycle. Benefits of pulmonary rehabilitation include decreased dyspnea, improved health-related quality of life, fewer days of hospitalization, and decreased health-care utilization.

As yet, there are no controlled studies on the use and effectiveness of pulmonary rehabilitation in the Indian setting and the optimum training regimen. This study aims to look at any improvements in the exercise capacity by means of objective incremental and field exercise tests, quality of life using validated questionnaires, severity of dyspnea, lung functions and nutritional parameters in patients who are diagnosed with severe forms of COPD after they have undergone a structured exercise training program.

Primary Objective • To assess the effect of structured outpatient pulmonary rehabilitation intervention on the six minute walk distance and health related quality of life in patients with chronic obstructive pulmonary disease.

Secondary Objectives

• To study the effects of pulmonary rehabilitation on:

* Maximum oxygen consumption (VO2max) and anaerobic threshold (AT)
* Lung functions: measured by changes in FEV1 and FVC
* Depression, Anxiety and Stress score (DASS)
* BODE (Body Mass Index, level of obstruction, level of dyspnea and exercise capacity) index
* Anthropometry: BMI and MUAC

Study design: Randomized Controlled Study Selection of subjects: Patients who have been diagnosed as Chronic Obstructive Pulmonary Disease visiting the outpatient clinic of the department of Pulmonary Medicine and Sleep Disorders Inclusion criteria

* Patients with severe COPD based on spirometry (FEV1 below 50%) presenting to pulmonary medicine outpatient clinic with modified medical research council (mMRC) grade 1 to 3.
* Those who are willing to participate in the study Exclusion criteria
* Patients on long term oxygen therapy or candidates for long term oxygen therapy
* Patients with severe orthopedic or neurological disorders limiting their mobility
* Exercise induced syncope
* Unstable angina or recent MI (within 4 months)
* Diagnosed Cognitive or active psychiatric disorders
* Comorbidities: uncontrolled hypertension >180/100
* Recent hospitalization for exacerbation within 6 weeks Sample size and location: 80 patients with diagnosed COPD presenting in the department of Pulmonary Medicine and Sleep Disorders, who will be randomized to 40 patients in each arm based on simple random sampling method.

Study Period: January 2015 to November 2017 Follow Up period: 8 weeks METHODOLOGY I. BASELINE EVALUATION After initial screening on patients with COPD in terms of severity, feasibility and commitment, patients who fulfill the inclusion and exclusion criteria will be randomized using computer generated random numbers to intervention and control groups. A baseline chest xray postero-anterior view (CXR-PA) view and a 12-lead electrocardiogram will be available before enrollment in the study. All patients will undergo pulmonary function test (PFT), cardiopulmonary exercise test using incremental cycle ergometry protocol (CPET), and six minute walk test (6MWT), along with the baseline demographic history and other relevant clinical information. CPET and 6MWT will be performed on two separate days. The six minute walking distance, VO2max and maximum work output during cycling and Saint George Respiratory Questionnaire will be recorded. Other nutritional parameters (mid-upper arm circumference, skin fold thickness), Depression Anxiety Stress Score, dyspnea scale and body mass index (BMI) will also be calculated and recorded. The 6MWT will be performed in accordance with the instructions of the American Thoracic Society, verbal encouragement will be given and the distance recorded. All these will be repeated at the end of 8 weeks. Tests will be separated by a minimum of one hour or until heart rate and oxygen saturation return to resting values.

II. RANDOMIZATION This will be done by using computer generated random numbers. III. EXERCISE TRAINING After the initial baseline evaluation, patients will be enrolled into the pulmonary rehabilitation program at the rehabilitation centre located in the premises of the department of pulmonary medicine and sleep disorders. The total duration of the program would be 12 weeks, with thrice weekly sessions of exercise training of minimum one hour duration. Participants will complete a minimum of 10 minutes each of treadmill walking, cycling, upper and lower limb resistance exercises at the 4 separated exercise stations located in the rehabilitation clinic of the Department of Pulmonary Medicine and Sleep Disorders. Rest period will be provided as required during the first 3 sessions. Second week onwards, participants will be encouraged to perform continuous training with intensity targeted at more than 60% of the maximum workload or till borg dyspnea scale of 4 to 6 is reached, with maximum of 10 minutes of rest per session during which breathing retraining exercises will be performed. It will then be followed by structured upper and lower limb strength exercises (e.g. sit-to-stand, foot treadling, thigh strengthening). Strength training will commence by performing one set of 8-12 repetitions of the exercise and progressed by increasing the number of sets from one to three gradually, targeting BORG dyspnea and fatigue scale of 4 to 6.

Adherence with training will be defined as completion of at least 80% of training sessions. All patients will be encouraged to perform daily activities such as walking and stair climbing and structured upper and lower limb exercises at home. (Manual/handouts provided). A diary will be provided to each of them to maintain daily symptoms and exercises at home.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe COPD based on spirometry (FEV1: <50%) presenting to pulmonary medicine outpatient clinic with mMRC grade 1 to 3.
* Those who are willing to participate in the study

Exclusion Criteria:

* Patients on long term oxygen therapy or candidates for long term oxygen therapy
* Patients with severe orthopedic or neurological disorders limiting their mobility
* Exercise induced syncope
* Unstable angina or recent MI (within 4 months)
* Diagnosed Cognitive or active psychiatric disorders
* Co morbidities: uncontrolled hypertension >180/100
* Recent hospitalization for exacerbation within 6 weeks

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To assess the change in health related quality of life in experimental arm (Saint George Respiratory Questionnaire) | 2 months
  Quality of life will be assessed by Saint George Respiratory Questionnaire
To assess the change in Six Minute Walk Distance in experimental arm | 2 months
  Exercise Capacity as measured by six minutes walk distance

SECONDARY OUTCOMES:
BODE index | 2 months
  The Index as calculated by body mass index (B), airway obstruction as measured by forced expiratory volume in one second (O), dyspnea grading (D) and exercise capacity (E)
Lung Functions | 2 months
  Lung functions as measured by spirometry that includes forced expiratory volume in one second (FEV1), forced vital capacity (FVC) and maximal inspiratory capacity.
Anxiety and Depression scale | 2 months
  The depression, anxiety and stress scale (DASS) will be used to assess the level of anxiety and depression in the subjects
Maximum exercise capacity | 2 months
  Cardiopulmonary exercise testing (CPET) will be used to assess change in maximum oxygen consumption and anaerobic threshold in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anant Mohan, MD, Study Director — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Science and Technology, Delhi, National Capital Territory of Delhi, India